CLINICAL TRIAL: NCT03778931
Title: Elacestrant Monotherapy vs. Standard of Care for the Treatment of Patients With ER+/HER2- Advanced Breast Cancer Following CDK4/6 Inhibitor Therapy: A Phase 3 Randomized, Open-label, Active-controlled, Multicenter Trial
Brief Title: Phase 3 Trial of Elacestrant Versus Standard of Care for the Treatment of ER+/HER2- Advanced Breast Cancer
Acronym: EMERALD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD1901-308
Record Dates: First submitted 2018-12-03; First posted 2018-12-19 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant; RAD1901; Standard of Care; Fulvestrant; Anastrozole; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elacestrant (Experimental): Participants in Arm 1 will receive elacestrant.
  Interventions: Drug: Elacestrant
- Standard of Care (SoC) (Active Comparator): Participants in Arm 2 will receive investigator's choice of one of the standard-of-care drugs (fulvestrant, anastrozole, letrozole, or exemestane).
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Elacestrant — 400 mg/day once daily oral dosing
  Other Names: RAD1901; ORSERDU
  Arms: Elacestrant
Drug: Standard of Care — * Fulvestrant: 500 mg administered intramuscularly (IM) into the buttocks as two 5 mL injections on C1D1, C1D15 and C2D1 and Day 1 of every subsequent 28-day cycle
  * Anastrozole 1 mg/day on a continuous dosing schedule
  * Letrozole: 2.5 mg/day on a continuous dosing schedule
  * Exemestane: 25 mg/day on a continuous dosing schedule
  Other Names: Faslodex, Arimidex, Femara, Aromasin
  Arms: Standard of Care (SoC)

SUMMARY:
This Phase 3 clinical study compares the efficacy and safety of elacestrant to the standard of care (SoC) options of fulvestrant or an aromatase inhibitor (AI) in women and men with breast cancer whose disease has advanced on at least one endocrine therapy including a CDK4/6 inhibitor in combination with fulvestrant or an aromatase inhibitor (AI).

DETAILED DESCRIPTION:
This is an international, multicenter, randomized, open-label, active-controlled, event-driven, Phase 3 clinical study comparing the efficacy and safety of elacestrant to the SoC options of fulvestrant or an aromatase inhibitor (AI) in postmenopausal women and in men with advanced or metastatic ER+/HER2- breast cancer, either in participants with tumors that harbor mutations in the ligand binding domain (LBD) of the estrogen receptor 1 (ESR1) gene (ESR1-mut participants) or in all participants regardless of ESR1 status (ESR1-mut and ESR1 wild type [ESR1-wt]) and whose disease has relapsed or progressed on at least one and no more than two prior lines of endocrine therapy (with documented progression), which must have included prior CDK4/6 inhibitor therapy in combination with fulvestrant or an aromatase inhibitor (AI) and for whom hormonal monotherapy with one of the SoC drugs (fulvestrant, anastrozole, letrozole, exemestane) is an appropriate treatment option.

ELIGIBILITY:
Critical Inclusion Criteria:

1. Participants with proven diagnosis of adenocarcinoma of the breast with evidence of either locally advanced disease not amenable to resection or radiation therapy with curative intent or metastatic disease not amenable to curative therapy.
2. Participants must be appropriate candidates for endocrine monotherapy
3. Participants must have measurable disease or bone only disease with evaluable lesions
4. Female or male participants age ≥ 18 years; female participants must be postmenopausal women, and male participants must not allow pregnancy with their sperm (abstain, do not donate sperm, et cetera).
5. Participants must have ER+ and HER2- tumor status
6. Participants must have previously received at least one and no more than two lines of endocrine therapy for advanced/metastatic breast cancer and meet additional previous treatment criteria.
7. Participants must have received prior treatment with a CDK4/6 inhibitor in combination with either fulvestrant or an aromatase inhibitor (AI) for advanced/metastatic breast cancer (mBC).
8. Participants may have received no more than one line of chemotherapy in the advanced/metastatic setting.

Critical Exclusion Criteria:

1. Prior treatment with elacestrant or other investigational selective estrogen receptor degrader (SERD) or ER antagonist (D-0502, GDC-0810, GDC-0927, GDC-9545, G1T-48, LSZ102, AZD9496, SAR439859, ZN-c5, H3B-6545, bazedoxifene, lasofoxifene).
2. Prior anticancer or investigational drug treatment within the following windows:

   1. Fulvestrant treatment < 42 days before first dose of study drug
   2. Any endocrine therapy < 14 days before first dose of study drug
   3. Chemotherapy < 21 days before first dose of study drug
   4. Any investigational anti-cancer drug therapy < 28 days or five half-lives (whichever is shorter) before the first dose of study drug. Enrollment of participants whose most recent therapy was an investigational agent should be discussed with the Sponsor
   5. Bisphosphonates or RANKL inhibitors initiated or dose changed < 3 months prior to first dose of study drug
3. Presence of symptomatic visceral disease as defined in protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (244):
- United States (104):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - St Bernard's Cancer Care, Jonesboro, Arkansas
  - St. Jude Heritage Healthcare, Fullerton, California
  - Adventist Health Glendale, Glendale, California
  - Moores Cancer Center at UC San Diego Health, La Jolla, California
  - Keck Hospital of USC-Norris Healthcare (HC3), Investigational Drug Service (IDS), Los Angeles, California
  - Keck Medical Center of USC, Los Angeles, California
  - USC IDS Pharmacy, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA West Medical Pharmacy 159, Los Angeles, California
  - TMPN Cancer Care, Redondo Beach, California
  - UC Davis Medical Center, Investigational Drug Service, Sacramento, California
  - UCSF Medical Center, San Francisco, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - Anschutz Cancer Center Pavilion, Aurora, Colorado
  - US Oncology - Rocky Mountain Cancer Centers - Midtown, Denver, Colorado
  - Poudre Valley Health Care, Inc. d/b/a Poudre Valley Health System, Fort Collins, Colorado
  - UCHealth Cancer Center, Fort Collins, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Piedmont Cancer Institute, P.C. - Oncology, Atlanta, Georgia
  - Suburban Hematology-Oncology Associates, Lawrenceville, Georgia
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Chicago Association for Research and Education in Science, Chicago, Illinois
  - Rush University Cancer Center, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Joliet Oncology-Hematology Associates, Joliet, Illinois
  - Presence Medical Group Hematology Oncology, Skokie, Illinois
  - Simmons Cancer Institute, Springfield, Illinois
  - Healthcare Research Network II, Tinley Park, Illinois
  - Fort Wayne Medical Oncology And Hematology, Fort Wayne, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Hematology Oncology Of Indiana, Indianapolis, Indiana
  - Cancer Resource Centre, Munster, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Pikeville Medical Center - Oncology/Hematology, Pikeville, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Highland Clinic, Shreveport, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - The Gynecologic Oncology Center at Mercy, Baltimore, Maryland
  - Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Maryland Oncology Hematology, Frederick, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Mass General Cancer Center at Newton Wellesley - Oncology, Boston, Massachusetts
  - Mass General North Shore Cancer Center - Oncology, Danvers, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Minnesota Oncology, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Jackson Oncology Associates, PLLC., Jackson, Mississippi
  - Chub O'Reilly Cancer Center, Springfield, Missouri
  - The Fred & Pamela Buffett Cancer Center, Omaha, Nebraska
  - Precision Cancer Research, Freehold, New Jersey
  - Saint Barnabas Medical Center - Cancer Center, Livingston, New Jersey
  - The Steeplechase Cancer Center, Somerville, New Jersey
  - New Mexico Oncology Hematology Consultants - Oncology, Albuquerque, New Mexico
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - New York Oncology Hematology, Albany, New York
  - Northern Westchester Hospital Cancer Center, Mount Kisco, New York
  - New York University Clinical Cancer Center, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Oncology and Hematology of White Plains, White Plains, New York
  - Carolina Institute For Clinical Research, Fayetteville, North Carolina
  - US Oncology Network, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Dayton Oncology & Hematology, Kettering, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Pinnacle Health Cancer Institute, Harrisburg, Pennsylvania
  - Abington Hematology Oncology Associates, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Charleston Oncology, Charleston, South Carolina
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - Brig Center For Cancer Care And Survivorship, Knoxville, Tennessee
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Austin Cancer Centers, Austin, Texas
  - Elligo Health Research, Austin, Texas
  - Texas Oncology-Beaumont, Beaumont, Texas
  - Texas Oncology-Methodist Dallas Cancer Center, Dallas, Texas
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Texas Oncology-Presbyterian Cancer Center Dallas, Dallas, Texas
  - Texas Oncology - Willowbrook, Houston, Texas
  - Texas Oncology - McAllen, McAllen, Texas
  - Texas Oncology-Mesquite, Mesquite, Texas
  - Texas Oncology-Paris, Paris, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Cancer Therapy and Research Center at UTHSCSA, San Antonio, Texas
  - Renovatio Medical The Woodlands, The Woodlands, Texas
  - Texas Oncology - The Woodlands, Gynecologic Oncology, The Woodlands, Texas
  - USO Texas Oncology - Tyler, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Fort Belvoir Community Hospital, Fort Belvoir, Virginia
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Colombia St. Mary's Medical Oncology, Milwaukee, Wisconsin
- Argentina (9):
  - Clínica Pergamino S.A., Pergamino, Buenos Aires
  - Fundacion CENIT para la Investigación en Neurociencias - Clinic, Buenos Aires, Buenos Aires F.D.
  - Oncología en Ciudad Autónoma de Buenos Aires, Buenos Aires, Buenos Aires F.D.
  - Centro Médico Austral, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - Oncología Médica, Rosario, Santa Fe Province
  - Clínica Caipo, San Miguel de Tucumán, Tucumán Province
  - Clínica Universitaria Reina Fabiola, Córdoba
  - Sanatorio del Salvador, Córdoba
  - Fundación CORI, La Rioja
- Australia (4):
  - Mater Misericordiae Ltd Mater Cancer Care Centre, Brisbane, Queensland
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Sunshine Coast University Hospital, Birtinya
  - Macarthur Cancer Therapy, Campbelltown
- Austria (5):
  - Department für Hämato-Onkologie - LKH Hochsteiermark, Leoben, Styria
  - Landeskrankenhaus (LKH) Leoben-Eisenerz, Leoben, Styria
  - Universitätsklinik Innsbruck, Innsbruck, Tyrol
  - Abteilung für Innere Medizin IV, Wels, Upper Austria
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria
- Belgium (19):
  - AZ Klina, Brasschaat, Antwerpen
  - UZ Antwerpen - Oncologie, Edegem, Antwerpen
  - AZ Turnhout, Turnhout, Antwerpen
  - Institut Jules Bordet - Oncologie Médicale, Brussels, Brussels Capital
  - CHU Brugmann, Brussels, Brussels Capital
  - UZ Brussel - Campus Jette, Brussels, Brussels Capital
  - Cliniques Universitaires Saint-Luc - Oncology, Brussels, Brussels Capital
  - Grand Hôpital de Charleroi - Site Notre-Dame, Charleroi, Hainaut
  - INDC Entité Jolimontoise - CH de Jolimont-Lobbes, Haine-Saint-Paul, Hainaut
  - Centre Hospitalier de l'Ardenne - Site de Libramont, Libramont, Luxembourg
  - Onze-Lieve-Vrouwziekenhuis Aalst, Aalst, Oost-Vlaanderen
  - AZ Nikolaas - Campus Sint-Niklaas Moerland, Sint-Niklaas, Oost-Vlaanderen
  - Universitaire Ziekenhuizen (UZ) - Leuven Cancer Institute, Leuven, Vlaams Brabant
  - AZ Sint-Jan Brugge - Oostende AV - Campus Sint-Jan - Oncology, Bruges, West-Vlaanderen
  - AZ Groeninge, Kortrijk, West-Vlaanderen
  - AZ Groeninge - Campus Kennedylaan, Kortrijk
  - CHU UCL Namur - Site Sainte-Elisabeth, Namur
  - CHU UCL Namur Campus Sainte-Elisabeth, Namur
  - Clinique Saint Pierre, Ottignies
- Canada (4):
  - Oncology and Haematology Clinic - Michael Garron Hospital, East York, Ontario
  - Pharmacie du CRCHUM, Montreal, Quebec
  - McGill University Health Centre - Cedars Cancer Center - Oncology, Montreal, Quebec
  - CHU de Quebec - Hopital du Saint Sacrement, Québec
- Denmark (5):
  - Vejle Sygehus, Vejle, Region Syddanmark
  - Næstved Sygehus, Næstved, Zeeland
  - Onkologisk Afdeling, Lillebælt Hospital, Vejle, Næstved, Zeeland
  - Aalborg Universitetshospital, Aalborg
  - Odense Universitetshospital - Oncology, Odense
- France (14):
  - Strasbourg Oncologie Libérale Centre de Radiothérapie, Strasbourg, Bas-Rhin
  - Centre de Lutte Contre le Cancer (CLCC), Caen, Calvados
  - IUCT-Oncopole Pharmacie-Essais Cliniques, Toulouse, Haute-Garonne
  - Hopital Trousseau - Service d'Oncologie Medicale, Tours, Indre-et-Loire
  - Centre Oscar Lambret, Department de Cancérologie Sénologique, Lille, Nord
  - Centre Jean Perrin, Clermont-Ferrand, Puy-de-Dôme
  - Centre Leon Berard Oncologie Médical, Lyon, Rhône
  - Hôpital Privé Jean Mermoz Département Pharmacie, Lyon, Rhône
  - Centre François Baclesse Service Pharmacie, Caen
  - Centre Georges Francois Leclerc, Dijon
  - Institut régional du Cancer Montpellier Service pharmacie-Essais cliniques, Montpellier
  - Centre DeLutte Contre Le Cancer - Institut Curie - Departement d'Oncologie Medica, Paris
  - Institut de Cancérologie Lucien Neuwirth Service pharmacie-Essais cliniques, Saint-Priest-en-Jarez
  - Institut Curie Saint-Cloud, Saint-Cloud, Île-de-France Region
- Greece (4):
  - University General Hospital Of Patras - Dpt Of Medicine, Division Oncology, Pátrai, Achaïa
  - Metropolitan Hospital - Oncology Unit, Athens, Attica
  - University General Hospital of Larissa, Larissa, Larisa
  - Bioclinic Thessaloniki, Thessaloniki
- Hungary (8):
  - Pécsi Tudományegyetem Klinikai Központ, Pécs, Baranya
  - Bács-Kiskun Megyei Kórház, Debrecen, Hajdú-Bihar
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz - Rendeloint, Szolnok, Jász-Nagykun-Szolnok
  - Szabolcs-Szatmár-Bereg Megyei Kórházak és Egyetemi Oktatókór, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Uzsoki Utcai Kórház, Budapest
  - Semmelweis Egyetem, Onkológiai Központ,, Budapest
  - Országos Onkológiai Intézet, Budapest
- Ireland (7):
  - Bon Secours Hospital [Oncology], Cork, Cork
  - Clinical Research Facility, St. James's Hospital, Dublin
  - Beaumont Hospital Cancer Clinical Trials Unit, Dublin
  - St Vincent's University Hospital, Dublin
  - Pharmacy Aseptic Compounding Unit Level 4, Sligo University Hospital, Sligo
  - Sligo University Hospital, Sligo
  - Pharmacy, UHW, Waterford
- Israel (9):
  - Sharett Institute of Oncology - Hadassah Medical Center, Jerusalem, Central District
  - The Chaim Sheba Medical Center, Tel-Hashomer, Central District
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah MO - Oncology, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center - Beilinson Hospital - Davidoff Cancer, Petah Tikva
  - Tel Aviv Sourasky Medical Center - Oncology, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (16):
  - Regional Cancer Center, Meldola, Forli-Cesena
  - IRCCS Istituto Clinico Humanitas Humanitas Cancer Center, Rozzano, Milano
  - Ospedale San Gerardo-ASST Monza, Monza, Monza E Brianza
  - Policlinico S.Orsola Malpighi, AOU di Bologna - SSD Oncol.Med. Addarii-Zamagni, Bologna
  - PO di Cremona, ASST di Cremona - Patologia Mammaria e Breast Unit - Cremona, Cremona
  - DiMI, Dipartimento di Medicina interna e Specialità mediche,, Genova
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - AOU Maggiore della Carità - SC Oncologia, Novara
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - IRCCS Policlinico San Matteo, Pavia
  - Via G. Dottore, 1 Sc Oncologia Medica Azienda Ospedaliera di Perugia, Perugia
  - SO S.Chiara, AOU Pisana - Oncologia 2, Pisa
  - Policlinico Universitario Campus Bio-medico, Università Campus Bio-medico di Roma,, Roma
  - Policlinico A. Gemelli, Roma
  - Azienda Sanitaria Universitaria Integrata di Udine, Udine
- Portugal (5):
  - Instituto Português de Oncologia de Coimbra, Coimbra
  - Hospital Senhora da Oliveira - Guimarães, E.P.E., Guimarães
  - Hospital da Luz, Lisbon
  - Instituto Português de Oncologia do Porto, Porto
  - Instituto Português Oncologia Francisco Gentil do Porto, Porto
- South Korea (8):
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - National Cancer Center, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (16):
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Universitario Son Espases, Servicio de Oncología, Palma de Mallorca, Balearic Islands
  - Hospital de Dia de Oncología, San Cristóbal de La Laguna, Canary Islands
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife, Canary Islands
  - Hospital Universitario de Fuenlabrada. Servicio de Oncología, Fuenlabrada, Madrid
  - Hospital de Navarra, Pamplona, Navarre
  - Hospital Xeral Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Clinic de Barcelona, Barcelona
  - M.D Anderson Center Madrid, Madrid
  - IOB Ruber Internacional, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Servicio de Oncología Médica Edificio Materno, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (7):
  - Mount Vernon Cancer Centre, Northwood, England
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Kent Oncology Centre, Maidstone Hospital, Maidstone, Kent
  - Taunton and Somerset NHS Trust, Taunton, Somerset
  - Velindre Cancer Centre - Oncology, Cardiff
  - University College London Hospitals, London
  - Sarah Cannon Research Institute, London

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Shah M, Lingam H, Gao X, Gittleman H, Fiero MH, Krol D, Biel N, Ricks TK, Fu W, Hamed S, Li F, Sun JJ, Fan J, Schuck R, Grimstein M, Tang L, Kalavar S, Abukhdeir A, Pathak A, Ghosh S, Bulatao I, Tilley A, Pierce WF, Mixter BD, Tang S, Pazdur R, Kluetz P, Amiri-Kordestani L. US Food and Drug Administration Approval Summary: Elacestrant for Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative, ESR1-Mutated Advanced or Metastatic Breast Cancer. J Clin Oncol. 2024 Apr 1;42(10):1193-1201. doi: 10.1200/JCO.23.02112. Epub 2024 Feb 21. PMID 38381994
- [Derived] Bidard FC, Kaklamani VG, Neven P, Streich G, Montero AJ, Forget F, Mouret-Reynier MA, Sohn JH, Taylor D, Harnden KK, Khong H, Kocsis J, Dalenc F, Dillon PM, Babu S, Waters S, Deleu I, Garcia Saenz JA, Bria E, Cazzaniga M, Lu J, Aftimos P, Cortes J, Liu S, Tonini G, Laurent D, Habboubi N, Conlan MG, Bardia A. Elacestrant (oral selective estrogen receptor degrader) Versus Standard Endocrine Therapy for Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: Results From the Randomized Phase III EMERALD Trial. J Clin Oncol. 2022 Oct 1;40(28):3246-3256. doi: 10.1200/JCO.22.00338. Epub 2022 May 18. Erratum In: J Clin Oncol. 2023 Aug 10;41(23):3962. doi: 10.1200/JCO.23.01239. PMID 35584336
- [Derived] Bardia A, Aftimos P, Bihani T, Anderson-Villaluz AT, Jung J, Conlan MG, Kaklamani VG. EMERALD: Phase III trial of elacestrant (RAD1901) vs endocrine therapy for previously treated ER+ advanced breast cancer. Future Oncol. 2019 Oct;15(28):3209-3218. doi: 10.2217/fon-2019-0370. Epub 2019 Aug 20. PMID 31426673

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SoC): Participants in Arm 2 will receive Investigator's choice of one of the standard-of-care drugs (fulvestrant, anastrozole, letrozole, or exemestane)
  Standard of Care:
  * Fulvestrant: 500 mg administered intramuscularly (IM) into the buttocks as two 5 mL injections on C1D1, C1D15 and C2D1 and Day 1 of every subsequent 28-day cycle
  * Anastrozole 1 mg/day on a continuous dosing schedule
  * Letrozole: 2.5 mg/day on a continuous dosing schedule
  * Exemestane: 25 mg/day on a continuous dosing schedule
Period: Overall Study
Arm/Group | Elacestrant | Standard of Care (SoC)
Started | 239 | 239
Intent-to-Treat Population | 239 | 239
Safety Population | 237 | 230
Completed (Only deaths indicated as leading to study discontinuation are reported in the Participant Flow section. All deaths regardless of causality or whether they were reported as a reason for study discontinuation are reported in the All-Cause Mortality section.) | 152 | 130 (Only deaths indicated as leading to study discontinuation are reported in the Participant Flow section. All deaths regardless of causality or whether they were reported as a reason for study discontinuation are reported in the All-Cause Mortality section.)
Not Completed | 87 | 109
Not completed — Withdrawal by Subject | 12 | 25
Not completed — Physician Decision | 1 | 3
Not completed — Participant Noncompliance | 1 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Death | 69 | 79

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elacestrant | Standard of Care (SoC) | Total
Number analyzed (Participants) | 239 | 239 | 478
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 135 | 128 | 263
  >=65 years | 104 | 111 | 215
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233 | 238 | 471
  Male | 6 | 1 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 18 | 37
  Not Hispanic or Latino | 194 | 191 | 385
  Unknown or Not Reported | 26 | 30 | 56
Height [Mean (Standard Deviation); unit: cm] — Population: Data was not collected for five participants
  cm
    number analyzed (Participants) | 236 | 237 | 473
    (all) | 162.27 (7.860) | 160.97 (7.149) | 161.62 (7.532)
Weight [Mean (Standard Deviation); unit: kg] | 72.70 (16.093) | 72.39 (16.390) | 72.55 (16.226)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Data was not collected for five participants
  kg/m^2
    number analyzed (Participants) | 236 | 237 | 473
    (all) | 27.58 (5.494) | 27.92 (5.853) | 27.75 (5.673)
Eastern Cooperative Oncology Group Performance Status [Count of Participants; unit: Participants] — Participants were graded on a scale from 0 to 5, where 5 was the worst:
  0. Normal activity. Fully active, able to carry on all pre-disease performance without restriction
  1. Symptoms, but ambulatory. Restricted in strenuous activity, ambulatory and able to carry out light work
  2. In bed <50% of time. Ambulatory, capable of all self-care, unable to carry out any work activities
  3. In bed >50% of time. Capable of limited self-care
  4. 100% bedridden. Completely disabled. Cannot carry out any self-care. Confined to bed or chair
  5. Dead
  Participants
    0: Fully active, able to carry on all pre-disease performance without restriction | 143 | 135 | 278
    1: Restricted in physically strenuous activity but ambulatory & can carry out light, sedentary work | 96 | 103 | 199
    2: Ambulatory and capable of all selfcare but unable to carry out any work activities | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival in ESR1-mut Participants
Description: Progression-free survival based on blinded IRC assessment in ESR1-mut participants defined as the length of time from randomization until the date of objective disease progression per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as assessed by the blinded IRC or death from any cause. Progression is defined per RECIST v1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From Date of Randomization until Disease Progression or Death Due to Any Cause (up to 12 Months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Elacestrant | Standard of Care (SoC)
Number analyzed (Participants) | 115 | 113
months | 3.78 [2.17 to 7.26] | 1.87 [1.87 to 2.14]
Statistical Analysis 1: Comparison: Elacestrant vs Standard of Care (SoC); The analysis was performed using a stratified Cox Proportional Hazards model with ties=Efron and the stratification factors: prior treatment with fulvestrant (yes vs no) and presence of visceral metastases (yes vs no); the CI calculated using a profile likelihood approach; Test type: Other; p = 0.0005, Log Rank; The p-value was generated by using a two-sided stratified log-rank test; Hazard Ratio (HR) = 0.546, 95% CI 2-sided [0.387 to 0.768]

2. Primary Outcome: Progression-free Survival in All Participants
Description: Progression-free survival based on blinded imaging review committee (IRC) assessment in all (ESR1-mut and ESR1-wt) participants.
Time Frame: From Date of Randomization until Disease Progression or Death Due to Any Cause (up to 12 Months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Elacestrant | Standard of Care (SoC)
Number analyzed (Participants) | 239 | 239
months | 2.79 [1.94 to 3.78] | 1.91 [1.87 to 2.10]
Statistical Analysis 1: Comparison: Elacestrant vs Standard of Care (SoC); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0018, Log Rank; The p-value was generated by using a two-sided stratified log-rank test; Hazard Ratio (HR) = 0.697, 95% CI 2-sided [0.552 to 0.880]

3. Secondary Outcome: Overall Survival in ESR1-mut Participants
Description: Overall survival in ESR1-mut participants, where overall survival is defined as the length of time from randomization until the date of death from any cause.
Time Frame: From Date of Randomization until Death Due to Any Cause (Estimated up to 24 Months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Elacestrant | Standard of Care (SoC)
Number analyzed (Participants) | 115 | 113
months | NA [18.60 to NA] — NA=not calculable (insufficient number of participants with events) | 16.95 [14.00 to NA] — NA=not calculable (insufficient number of participants with events)
Statistical Analysis 1: Comparison: Elacestrant vs Standard of Care (SoC); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.0325, Log Rank — The p-value was generated by using a two-sided stratified log-rank test; Hazard Ratio (HR) = 0.592, 95% CI 2-sided [0.361 to 0.958]

4. Secondary Outcome: Overall Survival in All Participants
Description: Overall survival in all (ESR1-mut and ESR1-wt) participants.
Time Frame: From Date of Randomization until Death Due to Any Cause (Estimated up to 24 Months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Elacestrant | Standard of Care (SoC)
Number analyzed (Participants) | 239 | 239
months | NA [19.29 to NA] — NA=not calculable (insufficient number of participants with events) | NA [15.80 to NA] — NA=not calculable (insufficient number of participants with events)
Statistical Analysis 1: Comparison: Elacestrant vs Standard of Care (SoC); Test type: Other; p = 0.0697, Log Rank; The p-value was generated by using a two-sided stratified log-rank test; Hazard Ratio (HR) = 0.742, 95% CI 2-sided [0.536 to 1.025] — Applied a stratified Cox Proportional Hazards model with ties=Efron and the stratification factors: ESR1-mutational status (ESR1-mut vs ESR1-wt), prior treatment with fulvestrant (yes vs no) and presence of visceral metastases (yes vs no)

ADVERSE EVENTS:
Time Frame: 24 months
Description: All-Cause Mortality, Progression-free Survival, and Overall Survival were assessed with the Intention-to-Treat Population, which consisted of all randomized participants. Adverse Events (Serious and Other) reporting reflects the Safety Population, which consisted of all participants who received at least 1 dose of study medication. All deaths regardless of causality are reported in the All-Cause Mortality section. Only deaths leading to study discontinuation are reported in the Participant Flow.
Arm/Group | Elacestrant | Standard of Care (SoC)
All-Cause Mortality (participants affected / at risk) | 70/239 | 80/239
Serious Adverse Events (participants affected / at risk) | 29/237 | 25/230
Other Adverse Events (participants affected / at risk) | 215/237 | 195/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elacestrant (N=237) | Standard of Care (SoC) (N=230)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 3
Septic shock (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spinal cord compression (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cranial nerve paralysis (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Meningeal disorder (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elacestrant (N=237) | Standard of Care (SoC) (N=230)
Anaemia (Blood and lymphatic system disorders) | 22 | 17
Nausea (Gastrointestinal disorders) | 83 | 44
Vomiting (Gastrointestinal disorders) | 45 | 20
Diarrhoea (Gastrointestinal disorders) | 33 | 22
Constipation (Gastrointestinal disorders) | 29 | 15
Dyspepsia (Gastrointestinal disorders) | 24 | 6
Abdominal pain (Gastrointestinal disorders) | 15 | 13
Fatigue (General disorders) | 45 | 44
Asthenia (General disorders) | 21 | 19
Injection site pain (General disorders) | 0 | 14
Urinary tract infection (Infections and infestations) | 16 | 12
Aspartate aminotransferase increased (Investigations) | 31 | 29
Alanine aminotransferase increased (Investigations) | 22 | 24
Blood alkaline phosphatase increased (Investigations) | 15 | 17
Decreased appetite (Metabolism and nutrition disorders) | 35 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 | 37
Back pain (Musculoskeletal and connective tissue disorders) | 32 | 22
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 14 | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 17
Headache (Nervous system disorders) | 29 | 26
Insomnia (Psychiatric disorders) | 18 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 12
Hot flush (Vascular disorders) | 27 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 14 | 15
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 12
Hypertension (Vascular disorders) | 9 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT03778931/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT03778931/SAP_003.pdf